CLINICAL TRIAL: NCT00201461
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate the Safety and Efficacy of the STARFlex® Septal Closure System Versus Best Medical Therapy in Patients With a Stroke and/or Transient Ischemic Attack Due to Presumed Paradoxical Embolism Through a Patent Foramen Ovale
Brief Title: Evaluation of the STARFlex® Septal Closure System in Patients With a Stroke or TIA Due to the Possible Passage of a Clot of Unknown Origin Through a Patent Foramen Ovale (PFO)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NMT Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G980031; CLOSURE I
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-11

CONDITIONS: Patent Foramen Ovale; Stroke; Ischemic Attack, Transient
Keywords: Patent Foramen Ovale; STARFlex; CLOSURE I; Septal Closure System; Stroke; Cerebrovascular Accident; Transient Ischemic Attack; Heart Septal Defects, Atrial
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke; Ischemic Attack, Transient; Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Best medical therapy
  Interventions: Drug: Best medical therapy
- 2 (Experimental): STARFlex arm
  Interventions: Device: STARFlex septal closure system

INTERVENTIONS:
Device: STARFlex septal closure system — transcatheter placement of STARFlex device to close a patent foramen ovale
  Arms: 2
Drug: Best medical therapy — aspirin (325 mg daily) and/or warfarin (target INR = 2.5)
  Arms: 1

SUMMARY:
The primary objective of the study is to determine whether the STARFlex® septal closure system will safely and effectively prevent a recurrent embolic stroke/transient ischemic attack (TIA) and mortality in patients with a PFO and to demonstrate superiority of the STARFlex® device compared to best medical therapy.

ELIGIBILITY:
Major Inclusion Criteria:

* Age 18-60 years inclusive.
* Positive contrast valsalva bubble study by trans-esophageal echocardiogram (TEE) for patent foramen ovale (PFO), with or without atrial septal aneurysm.
* Stroke or clinically definite TIA (contact study coordinator).
* Be able to comply with follow up over two years.
* Be competent to, or have a legal guardian competent to, provide informed consent following full disclosure of risks and benefits of both treatment arms by a study investigator.
* Venous access capable of accepting a 10F minimum vascular sheath.
* Have, or be willing to, discontinue hormonal based contraceptive use prior to enrollment and for the term of the study.
* Has cardiac anatomy based on enrollment echocardiogram that will allow for placement of the implant if randomized to the implant arm.
* Note: Additional inclusion criteria may apply. Contact study coordinator or principal investigator for details.

Post-randomization - device patients only

* The size of the PFO (measured by indentation with a soft balloon) must be amenable to selection of a STARFlex device.

Major Exclusion Criteria:

* Carotid artery stenosis > 50%.
* Intracranial stenosis > 50% appropriate to symptoms.
* Complex aortic arch atheroma with high risk features for embolism
* Aortic arch, carotid or vertebral artery dissection.
* Mitral or aortic valve stenosis, vegetation, or calcification > 5 mm mitral annular calcification (MAC) thickness.
* Active pregnancy.
* Active infections (contact study coordinator).
* Active infective endocarditis or bacteremia.
* Prosthetic heart valves in any location.
* Anterior MI within 3 months of neurological event.
* Chronic atrial fibrillation
* Thrombus in, or occluded, venous access route.
* Contraindication to heparin, aspirin, clopidogrel, or warfarin, or a known medical condition that requires continuous warfarin.
* Patient enrolled in another investigation study where clinical endpoint interference may occur.
* Permanent pacemaker or inferior vena cava (IVC) filter.
* Serum creatinine > 2.0 mg/dL
* Patients with known vasculitis or neurologic disorder.
* Baseline modified Rankin score of 3 or more.
* Hypercoagulopathies requiring long-term warfarin.
* Note: Additional exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2003-06; Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Two (2) year incidence of stroke or Hard TIA | 2 years
All cause mortality for the first 30 days of follow up/discharge, whichever is longer | 30 days
Neurological mortality from 31 days of follow up (F/U) or longer | 31 days

SECONDARY OUTCOMES:
Incidence of primary endpoint as a total and broken down by event type/treatment group in: stroke/TIA patients (pts) and DW-MR+ pts with symptoms < 24 hours | < 24 hrs
Incidence of primary endpoint in BMT group | 2 years
Per treatment group, incidence of relevant/notable adverse events (AEs) | 2 years
Device group: (1) Incidence of primary endpoint in pts prescribed aspirin (325 versus 81 mg) daily, (2) Incidence of relevant/notable AEs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Furlan, MD, Principal Investigator — Cleveland Clinic Foundation, Cleveland, OH; Mark Reisman, MD, Principal Investigator — Swedish Medical Center, Seattle, WA
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Elmariah S, Furlan AJ, Reisman M, Burke D, Vardi M, Wimmer NJ, Ling S, Chen X, Kent DM, Massaro J, Mauri L; CLOSURE I Investigators. Predictors of recurrent events in patients with cryptogenic stroke and patent foramen ovale within the CLOSURE I (Evaluation of the STARFlex Septal Closure System in Patients With a Stroke and/or Transient Ischemic Attack Due to Presumed Paradoxical Embolism Through a Patent Foramen Ovale) trial. JACC Cardiovasc Interv. 2014 Aug;7(8):913-20. doi: 10.1016/j.jcin.2014.01.170. PMID 25147037
- [Derived] Furlan AJ, Reisman M, Massaro J, Mauri L, Adams H, Albers GW, Felberg R, Herrmann H, Kar S, Landzberg M, Raizner A, Wechsler L; CLOSURE I Investigators. Closure or medical therapy for cryptogenic stroke with patent foramen ovale. N Engl J Med. 2012 Mar 15;366(11):991-9. doi: 10.1056/NEJMoa1009639. PMID 22417252
- [Derived] Furlan AJ, Reisman M, Massaro J, Mauri L, Adams H, Albers GW, Felberg R, Herrmann H, Kar S, Landzberg M, Raizner A, Wechsler L; CLOSURE I Investigators. Study design of the CLOSURE I Trial: a prospective, multicenter, randomized, controlled trial to evaluate the safety and efficacy of the STARFlex septal closure system versus best medical therapy in patients with stroke or transient ischemic attack due to presumed paradoxical embolism through a patent foramen ovale. Stroke. 2010 Dec;41(12):2872-83. doi: 10.1161/STROKEAHA.110.593376. Epub 2010 Nov 4. PMID 21051670